CLINICAL TRIAL: NCT00546819
Title: A Phase IIb Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of Zoster Vaccine Live (Oka/Merck) in Patients on Chronic/Maintenance Corticosteroids
Brief Title: ZOSTAVAX™ in Patients on Chronic/Maintenance Corticosteroids (V211-017) (COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-017; 2006_557
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ZOSTAVAX™ (Experimental): Participants administered ZOSTAVAX™ on Day 1.
  Interventions: Biological: Zoster Vaccine, Live
- Placebo (Placebo Comparator): Participants administered Placebo on Day 1.
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Zoster Vaccine, Live — A single dose of 0.65 ml Zoster Vaccine, Live, injected subcutaneously on Day 1
  Other Names: V211
  Arms: ZOSTAVAX™
Biological: Comparator: Placebo — A single dose of 0.65 ml Placebo to ZOSTAVAX™ injected subcutaneously on Day 1.
  Arms: Placebo

SUMMARY:
The purpose of the study was to assess the safety, tolerability, and immunogenicity of ZOSTAVAX™ in patients receiving chronic/maintenance corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Varicella-history positive, herpes zoster (HZ)-history negative patients
* 60 years of age and older receiving chronic/maintenance systemic corticosteroid therapy at a daily dose of 5 to 20 mg of prednisone or equivalent for at least the 2 weeks immediately prior to enrollment and expected to continue to receive a daily dose of 5 to 20 mg of prednisone or equivalent for the 6-week primary safety follow-up period (dose may vary within this range during the 6-week postvaccination period)
* All females enrolling must be postmenopausal

Exclusion Criteria:

* Patients with a history of hypersensitivity reaction to gelatin or neomycin
* Prior receipt of varicella or zoster vaccine; prior history of herpes zoster
* Immune globulin and/or blood products given within 5 months prior to or expected within the 6-week postvaccination period
* Receipt of any live virus vaccinations within 1 month or receipt of any inactivated vaccinations within 7 days prior to enrollment
* Known immune deficiency that is caused by a medical condition
* Any use in the 8 weeks prior to vaccination or for 6 weeks after vaccination other medications which may suppress the immune system including methotrexate, corticosteroids at a daily dose greater than 20 mg of prednisone or equivalent, agents used to treat cancer, or medications which alter the level of the immune response used to treat arthritis or other illnesses
* Concomitant use of antiviral therapy
* A history of alcohol abuse or recreational drug use

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Russell AF, Parrino J, Fisher CL Jr, Spieler W, Stek JE, Coll KE, Su SC, Xu J, Li X, Schlienger K, Silber JL. Safety, tolerability, and immunogenicity of zoster vaccine in subjects on chronic/maintenance corticosteroids. Vaccine. 2015 Jun 17;33(27):3129-34. doi: 10.1016/j.vaccine.2015.04.090. Epub 2015 May 8. PMID 25964168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ZOSTAVAX™ | Placebo
Started | 207 | 102
VACCINATED | 206 | 100
Completed | 199 | 96
Not Completed | 8 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX™ | Placebo | Total
Number analyzed (Participants) | 207 | 102 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (6.9) | 69.9 (7.2) | 69.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 80 | 220
  Male | 67 | 22 | 89
Daily Corticosteroid Dose Stratum [Number; unit: Participants]
  5 to 10 mg of prednisone or equivalent | 182 | 88 | 270
  >10 to 20 mg of prednisone or equivalent | 25 | 14 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: A serious adverse event is defined as any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement.
Time Frame: Up to 182 days postvaccination
Population: All participants who were vaccinated and had any safety
  follow-up were included in the safety analysis.
Measure: Number; unit: Participants
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 204 | 99
Participants | 21 | 11

2. Secondary Outcome: Geometric Mean Titer (GMT) of Varicella-Zoster Virus (VZV) Antibodies at 42 Days Postvaccination
Description: The Geometric Mean Titer (GMT) of VZV antibodies in participants' serum samples was assessed by a glycoprotein enzyme-linked immunosorbent assay (gpELISA).
Time Frame: 42 days postvaccination
Population: Per-protocol population: All vaccinated participants who had serology results and who had no protocol deviations that would interfere with the evaluation of VZV-specific gpELISA antibody response.
Measure: Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 167 | 88
gpELISA units/mL | 531.1 [453.3 to 622.1] | 224.3 [169.8 to 296.2]

3. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of the VZV Antibody Response From Day 1 to Day 42 Postvaccination.
Description: The geometric mean fold rise (GMFR) of the VZV antibodies from Day 1 to Week 6 postvaccination.
Time Frame: 42 days postvaccination
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 167 | 88
Ratio | 2.3 [2.0 to 2.7] | 1.1 [1.0 to 1.2]

ADVERSE EVENTS:
Time Frame: Up to 182 days postvaccination for serious adverse events and 42 days postvaccination for other adverse events.
Arm/Group | ZOSTAVAX™ | Placebo
Serious Adverse Events (participants affected / at risk) | 21/204 | 11/99
Other Adverse Events (participants affected / at risk) | 43/204 | 10/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX™ (N=204) | Placebo (N=99)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZOSTAVAX™ (N=204) | Placebo (N=99)
Injection site erythema (General disorders) | 36 (39) | 4 (4)
Injection site pain (General disorders) | 22 (23) | 8 (8)
Injection site swelling (General disorders) | 23 (24) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. SPONSOR review can be expedited to meet publication guidelines.